CLINICAL TRIAL: NCT01006395
Title: Prevention of Micro-architectural Bone Decay in Males With Non-metastatic Prostate Cancer Receiving Androgen Deprivation Therapy (ADT)
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Austin Health (Other Government)
Responsible Party: Principal Investigator, Mathis Grossmann, Associate Prof, Austin Health
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MG2009_01
Record Dates: First submitted 2009-11-01; First posted 2009-11-02 (Estimated); Last update posted 2019-07-05 (Actual); Status verified 2019-07

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; Androgen deprivation; Bone Health; Insulin resistance; Men with nonmetastatic prostate cancer receiving androgen deprivation
MeSH Terms: conditions — Prostatic Neoplasms; Insulin Resistance | interventions — Zoledronic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- zoledronic acid (Active Comparator): intervention
  Interventions: Drug: Zoledronic acid
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Zoledronic acid — yearly infusion
  Arms: zoledronic acid
Drug: Placebo — yearly infusion
  Arms: Placebo

SUMMARY:
Less than 20% of men in whom prostate cancer is diagnosed early die from it. Cardiovascular disease is the most common cause of death in men with early prostate cancer. A commonly used form of treatment for prostate cancer is androgen deprivation therapy (ADT). ADT, while effective for the treatment of prostate cancer, has been linked to undesirable side effects, such as an increased risk of bone fractures and diabetes. Bisphosphonates, a class of drugs that prevent bone resorption, have been show to reduce the loss of bone mineral density that occurs as a consequence of ADT, but the effects of bisphosphonates on preservation of bone architecture is unknown.

This project has two main goals:

To assess prospectively, in men with prostate cancer receiving ADT, the effect of:

1. the intravenous bisphosphonate zoledronic acidon ADT-induced microarchitectural decay of bone structure.
2. ADT on insulin resistance and glucose metabolism. We will recruit 100 ambulatory men with non-metastatic prostate cancer who are about to commence a three year course of ADT as per routine clinical practice at Austin Health. Men will be randomised to receive either intravenous zoledronic acid (Aclasta, Novartis Pharmaceuticals) or placebo at baseline and after 12 months of ADT. Men with contraindications to zoledronic acid will be excluded from the study. All 100 study subjects will have clinical and laboratory assessment at baseline, and at 3, 6, 12, 18 and 24 months (study end), and imaging studies at baseline and at 6, 12 and 24 months.

The study protocol is outlined in more detail below (Please see flow chart included in the in

PICF):

Clinical and laboratory assessment:

Full medical history, physical examination and quality of life assessment using the SF-36 questionnaire. Laboratory studies will include: oral glucose tolerance test (3, 12 and 24 months Commercial-in-Confidence only) and measurements of measure total testosterone, fasting glucose, C-peptide, HBA1c, bone turnover markers.

Imaging studies:

1. Bony micro-architecture by high resolution quantitative computed tomography
2. Bone mineral density and body composition by DEXA This project will have no direct benefit for the subjects involved in this study; however, it will improve our understanding on the effect of zoledronic acid on bone microarchitecture in men with prostate cancer receiving ADT. It will also help us to better understand the effect of ADT on insulin resistance and glucose metabolism.

DETAILED DESCRIPTION:
Not desired

ELIGIBILITY:
Inclusion Criteria:

* Men with prostate cancer receiving ADT

Exclusion Criteria:

* Contraindications to Zoledronic acid

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2011-01; Primary Completion 2019-04 (Actual); Study Completion 2019-04 (Actual)

PRIMARY OUTCOMES:
Bone microarchitecture | 24 months

SECONDARY OUTCOMES:
Insulin resistance | 24 months

CONTACTS AND LOCATIONS:
Locations (1):
- Austin Health, Heidelberg, Victoria, Australia

REFERENCES:
- [Derived] Cheung AS, Hoermann R, Zhu J, Lim Joon D, Zajac JD, Grossmann M. Zoledronic acid does not affect insulin resistance in men receiving androgen deprivation therapy: a prespecified secondary analysis of a randomised controlled trial. Ther Adv Endocrinol Metab. 2021 May 5;12:20420188211012118. doi: 10.1177/20420188211012118. eCollection 2021. PMID 34104395